CLINICAL TRIAL: NCT01332838
Title: A Comparison of Specialized Versus Standard Compression After Saphenous Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Washington (Other)
Collaborators: Lake Washington Vascular (Other); Sigvaris, Inc (Unknown)
Responsible Party: Mark Meissner, MD, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COSSCA
Record Dates: First submitted 2011-03-30; First posted 2011-04-11 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Stockings, Compression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Sigvaris special compression stocking (Experimental)
  Interventions: Device: compression stockings (Sigvaris )
- Standard Compression (Active Comparator)
  Interventions: Procedure: Compression stockings

INTERVENTIONS:
Procedure: Compression stockings — standard 30to 40 mm Hg thigh high compression stockings
  Arms: Standard Compression
Device: compression stockings (Sigvaris ) — Specialized monoleg compression
  Arms: Sigvaris special compression stocking

SUMMARY:
The purpose of this study is to determine if the use of specialized compression garments, in comparison to standard compression, improves early patient outcomes after endovenous ablation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* CEAP Class C2 or C3 disease
* Incompetence of the great saphenous vein defined a reflux persisting>0.5 seconds in the upright position
* Planned endovenous ablation of the great saphenous vein

Exclusion Criteria:

* Inability of patient or legal guardian to provide informed consent
* Previous history of DVT
* Clinical evidence of significant chronic venous disease (CEAP classes C4, C5, C6)
* Planned concomitant phlebectomy or sclerotherapy within 4 weeks of endovenous ablation
* Documented allergy or intolerance to compression stockings
* Arterial insufficiency as documented by an ankle-brachial index <0.5
* Known prothrombotic condition
* Life expectancy less than 1 year
* Inability to return for follow-up due to geographic inaccessibility, concurrent medical conditions or substance abuse
* Weight greater than 220 pounds or height > 6'4"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Behavioral Recovery After Varicose Veins (BRAVV) score. | 7 days

SECONDARY OUTCOMES:
Additional scoring and venous duplex ultrasonography | 7 and 28 days
  Behavioral Recovery After Varicose Veins (BRAVV) score at 28 days, Pain score at 7 and 28 days, Bruising score at 7 and 28 days, Venous Clinical Severity Score (VCSS) at 7 and 28 days, venous duplex ultrasonography at 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States